CLINICAL TRIAL: NCT04353063
Title: Assessment and Management of Muscle Wasting in Children and Adolescents With Cancer
Brief Title: Muscle Wasting in Children and Adolescents With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202001023RINA
Record Dates: First submitted 2020-04-08; First posted 2020-04-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-03

CONDITIONS: Cachexia; Cancer; Muscle Wasting; Child Development; Adolescent Development
Keywords: symptom distress; nutrition; physical activity; body composition; children and adolescents; cancer; nursing care
MeSH Terms: conditions — Cachexia; Neoplasms; Muscular Atrophy; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The patients in the control group will not receive any walking exercise education until the 4-week intervention ends. They will then receive the same education material ("How walking is beneficial to your health") and will be told about the benefits of walking.
- experimental group (Experimental): Participants in the experimental group will also be educated on the general use of the ActiGraph through verbal and written information and will be asked to wear the ActiGraph during week 0 for 3 consecutive days. The collected physical activity parameters will be the baseline data.Afterward, participants in the experimental group will be educated with the educational materials "How walking is beneficial to muscle mass and your health." And then the ActiGraph will be collected by the research assistant in order to analyze the physical activity parameters, including time spent walking and walking steps. A final assessment will be conducted at week 4. The participant will be reminded that the ActiGraph and the post-test questionnaires will be picked up at the end of week 4.
  Interventions: Behavioral: Multidisciplinary care with a personalized care

INTERVENTIONS:
Behavioral: Multidisciplinary care with a personalized care — During the 4-week intervention, participants will be given stickers by the research assistant to increase their motivation to walk. A sticker will be given once a participant reaches a daily walking-time goal. The number of stickers participants receive depends on the number of days they reach their daily goals. The stickers can be redeemed for the participant's choice of gift in the gift shelf of the ward or on a gift card. A final assessment will be conducted at week 4. The participant will be reminded that the ActiGraph and the post-test questionnaires will be picked up at the end of week 4
  Arms: experimental group

SUMMARY:
The series of the 3-year study aims to explore parents' experience of caring for a child's weight change among parents of children and adolescents with cancer, examine the associations and trends among muscle wasting and health-related variables, and then implement and assess effectiveness of a multidisciplinary approach with a personalized physical activity (walking) training intervention on improving muscle mass and other health-related variables.

DETAILED DESCRIPTION:
Specific aims, year by year

1. The aim for Year 1 is as follows:

   Aim 1: To explore parents' experience of caring for promoting a child's exercise among parents of children and adolescents with cancer.
2. The aims for Year 2 are as follows:

   Aim 2-1: To examine the associations between the degree of muscle wasting and health-related variables (fatigue level, symptom distress level, physical activity involvement, dietary intake, and QoL) among children and adolescents with cancer.

   Aim 2-2: To examine the trends of changes in muscle wasting and health-related variables (fatigue level, symptom distress level, physical activity involvement, dietary intake, and QoL) during the first 6 months of cancer treatment among children and adolescents with cancer.
3. The aim for Year 3 is as follows:

Aim 3: To examine the effectiveness of a multidisciplinary approach with a personalized walking exercise program on changes in body composition and health-related variables (fatigue level, symptom distress level, subjective physical activity involvement, objective physical activity measurement, dietary intake, and QoL) among children and adolescents with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1:(1) parents of children diagnosed with malignancies at 3-18 years old, (2) whose children have received cancer treatment for at least 6 months, (3) who are the main caregivers, and (4) who are willing to participate in the study.
* Aim 2-1:(1) children and adolescents diagnosed with malignancies at 3-18 years old, (2) who are previously or currently treated for cancer, and (3) who are willing to participate in the study. Two hundred patients will be recruited.
* Aim 2-2:(1) children and adolescents diagnosed with malignancies at 3-18 years old, (2) newly diagnosed with cancer within the past 1 month, and (3) willing to participate in the study. One hundred participants will be recruited.
* Aim 3:(1) children and adolescents aged 3-18 years old and are undergoing treatment, and (2) who are willing to participate in the study.

Exclusion Criteria:

-Aim 1-3: Children and adolescents are under poor physical or cognitive conditions.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 440 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Demographics | baseline
  age, age at diagnosis, diagnosis, cancer recurrence or not, treatment status, gender, education, parents' education, height, and body weight.
Lab data | baseline
  protein profile (albumin), lipid profile (TG, cholesterol, LDH, HDH), liver profile (GOT, GPT), CBC profile (HB, RBC, WBC/DC, platelet), renal profile (BUN, CRE), inflammation index (CRP), and sugar profile (Glucose-AC and HbA1C) at diagnosis and at study baseline.
Medication dosage | baseline
  accumulated corticosteroid dosage, accumulated radiation dosage.
Cachexia assessment | baseline
  This assessment includes weight loss grading and muscle power grading. Weight loss grading uses a 5x5 matrix to grade the patient's level of cancer-associated weight loss.Grade 0 = complete paralysis; Grade 1 = flicker of contraction present; Grade 2 = active movement with gravity eliminated; Grade 3 = active movement against gravity; Grade 4 = active movement against gravity and some resistance described as poor, fair, or moderate strength; and Grade 5 = normal power.
Inbody S10 | Week 0
  The InBody S10 BIA device measures resistance at six frequencies (1, 5, 50, 250, 500, and 1000 KHz).
Inbody S10 | Week 4
  The InBody S10 BIA device measures resistance at six frequencies (1, 5, 50, 250, 500, and 1000 KHz).
Multidimensional Fatigue Scale (MFS): | week 4
  MFS versions are designed for ages 5-18. The parent proxy reports, which include children 2-4 years of age (toddler), are used to assess the parent's perception of their child's fatigue. The instrument consists of 18 items. Patients are assessed on how often a particular problem occurred in the past month by using a 5-point Likert scale from 0 to 4 and rescaled to 0-100, so that higher scores indicate fewer symptoms of fatigue.
Symptom Distress Scale (SDS) | Week 0(baseline)
  The SDS is a 5-point mixed-response scale with 13 items that measure symptom distress. Total scores range from 13 to 65; higher scores indicate more severe symptom distress during the past week.
Symptom Distress Scale (SDS) | week 1
  The SDS is a 5-point mixed-response scale with 13 items that measure symptom distress. Total scores range from 13 to 65; higher scores indicate more severe symptom distress during the past week.
Symptom Distress Scale (SDS) | week 2
  The SDS is a 5-point mixed-response scale with 13 items that measure symptom distress. Total scores range from 13 to 65; higher scores indicate more severe symptom distress during the past week.
Symptom Distress Scale (SDS) | week 3
  The SDS is a 5-point mixed-response scale with 13 items that measure symptom distress. Total scores range from 13 to 65; higher scores indicate more severe symptom distress during the past week.
Symptom Distress Scale (SDS) | week 4
  The SDS is a 5-point mixed-response scale with 13 items that measure symptom distress. Total scores range from 13 to 65; higher scores indicate more severe symptom distress during the past week.
Exercise Involvement Scale (EIS) | Week 0(baseline)
  Exercise involvement is calculated by the equation: Exercise Involvement Score = exercise frequency x (exercise intensity + exercise duration). The total score represents an individual's level of exercise involvement. There are six graded response options, ranging from 1 (zero) to 6 (5 or more times a week). A higher score indicates more frequent exercise during the past week.
Exercise Involvement Scale (EIS) | week 1
  Exercise involvement is calculated by the equation: Exercise Involvement Score = exercise frequency x (exercise intensity + exercise duration). The total score represents an individual's level of exercise involvement. There are six graded response options, ranging from 1 (zero) to 6 (5 or more times a week). A higher score indicates more frequent exercise during the past week.
Exercise Involvement Scale (EIS) | week 2
  Exercise involvement is calculated by the equation: Exercise Involvement Score = exercise frequency x (exercise intensity + exercise duration). The total score represents an individual's level of exercise involvement. There are six graded response options, ranging from 1 (zero) to 6 (5 or more times a week). A higher score indicates more frequent exercise during the past week.
Exercise Involvement Scale (EIS) | week 3
  Exercise involvement is calculated by the equation: Exercise Involvement Score = exercise frequency x (exercise intensity + exercise duration). The total score represents an individual's level of exercise involvement. There are six graded response options, ranging from 1 (zero) to 6 (5 or more times a week). A higher score indicates more frequent exercise during the past week.
Exercise Involvement Scale (EIS) | week 4
  Exercise involvement is calculated by the equation: Exercise Involvement Score = exercise frequency x (exercise intensity + exercise duration). The total score represents an individual's level of exercise involvement. There are six graded response options, ranging from 1 (zero) to 6 (5 or more times a week). A higher score indicates more frequent exercise during the past week.
Visual analogue scale for dietary intake (VAS-DI) | Week 0(baseline)
  Patients are asked to answer the question: "If you consider that, at times when you are in good health, you eat 10 out of 10, how much do you currently eat on a scale from 0 to 10?" A response of 0 would mean eating "nothing at all" and 10 would be eating "as usual." For patients who do not understand this question, the researcher helps by adding: "How do you currently eat at this moment: a quarter of the usual amount, half of the usual amount, or three-quarters of the usual amount?" Patients tick a 100-mm line traced on paper to answer the inquiry "How much do you currently eat on a scale from 0 'nothing' (far left side of the line) to 10 'as usual' (far right side of the line)?" The left extremity of the line is anchored by "I eat nothing at all" (0 cm), the middle by "I eat half the usual amount" (5 cm), and the right extremity by "I eat as usual" (10 cm).
Visual analogue scale for dietary intake (VAS-DI) | week 1
  Patients are asked to answer the question: "If you consider that, at times when you are in good health, you eat 10 out of 10, how much do you currently eat on a scale from 0 to 10?" A response of 0 would mean eating "nothing at all" and 10 would be eating "as usual." For patients who do not understand this question, the researcher helps by adding: "How do you currently eat at this moment: a quarter of the usual amount, half of the usual amount, or three-quarters of the usual amount?" Patients tick a 100-mm line traced on paper to answer the inquiry "How much do you currently eat on a scale from 0 'nothing' (far left side of the line) to 10 'as usual' (far right side of the line)?" The left extremity of the line is anchored by "I eat nothing at all" (0 cm), the middle by "I eat half the usual amount" (5 cm), and the right extremity by "I eat as usual" (10 cm).
Visual analogue scale for dietary intake (VAS-DI) | week 2
  Patients are asked to answer the question: "If you consider that, at times when you are in good health, you eat 10 out of 10, how much do you currently eat on a scale from 0 to 10?" A response of 0 would mean eating "nothing at all" and 10 would be eating "as usual." For patients who do not understand this question, the researcher helps by adding: "How do you currently eat at this moment: a quarter of the usual amount, half of the usual amount, or three-quarters of the usual amount?" Patients tick a 100-mm line traced on paper to answer the inquiry "How much do you currently eat on a scale from 0 'nothing' (far left side of the line) to 10 'as usual' (far right side of the line)?" The left extremity of the line is anchored by "I eat nothing at all" (0 cm), the middle by "I eat half the usual amount" (5 cm), and the right extremity by "I eat as usual" (10 cm).
Visual analogue scale for dietary intake (VAS-DI) | week 3
  Patients are asked to answer the question: "If you consider that, at times when you are in good health, you eat 10 out of 10, how much do you currently eat on a scale from 0 to 10?" A response of 0 would mean eating "nothing at all" and 10 would be eating "as usual." For patients who do not understand this question, the researcher helps by adding: "How do you currently eat at this moment: a quarter of the usual amount, half of the usual amount, or three-quarters of the usual amount?" Patients tick a 100-mm line traced on paper to answer the inquiry "How much do you currently eat on a scale from 0 'nothing' (far left side of the line) to 10 'as usual' (far right side of the line)?" The left extremity of the line is anchored by "I eat nothing at all" (0 cm), the middle by "I eat half the usual amount" (5 cm), and the right extremity by "I eat as usual" (10 cm).
Visual analogue scale for dietary intake (VAS-DI) | week 4
  Patients are asked to answer the question: "If you consider that, at times when you are in good health, you eat 10 out of 10, how much do you currently eat on a scale from 0 to 10?" A response of 0 would mean eating "nothing at all" and 10 would be eating "as usual." For patients who do not understand this question, the researcher helps by adding: "How do you currently eat at this moment: a quarter of the usual amount, half of the usual amount, or three-quarters of the usual amount?" Patients tick a 100-mm line traced on paper to answer the inquiry "How much do you currently eat on a scale from 0 'nothing' (far left side of the line) to 10 'as usual' (far right side of the line)?" The left extremity of the line is anchored by "I eat nothing at all" (0 cm), the middle by "I eat half the usual amount" (5 cm), and the right extremity by "I eat as usual" (10 cm).
PedsQL | Week 0(baseline)
  The PedsQL Cancer Module is designed to measure pediatric cancer-specific health-related QoL in patients ages 2-18 years. The scale consists of 27 items that address eight dimensions: pain and hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance, and communication. Items are rated on a 5-point scale
PedsQL | week 4
  The PedsQL Cancer Module is designed to measure pediatric cancer-specific health-related QoL in patients ages 2-18 years. The scale consists of 27 items that address eight dimensions: pain and hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance, and communication. Items are rated on a 5-point scale
ActiGraph | Week 0(baseline)
  The ActiGraph GT3X accelerometer is a reliable and valid tool for assessing objective activity level, validated in participants ages 7-18 years. It captures and records continuous raw acceleration data, which will be downloaded in 60-second epochs using ActiLife 6.13.3 software.
ActiGraph | week 1
  The ActiGraph GT3X accelerometer is a reliable and valid tool for assessing objective activity level, validated in participants ages 7-18 years. It captures and records continuous raw acceleration data, which will be downloaded in 60-second epochs using ActiLife 6.13.3 software.
ActiGraph | week 2
  The ActiGraph GT3X accelerometer is a reliable and valid tool for assessing objective activity level, validated in participants ages 7-18 years. It captures and records continuous raw acceleration data, which will be downloaded in 60-second epochs using ActiLife 6.13.3 software.
ActiGraph | week 3
  The ActiGraph GT3X accelerometer is a reliable and valid tool for assessing objective activity level, validated in participants ages 7-18 years. It captures and records continuous raw acceleration data, which will be downloaded in 60-second epochs using ActiLife 6.13.3 software.
ActiGraph | week 4
  The ActiGraph GT3X accelerometer is a reliable and valid tool for assessing objective activity level, validated in participants ages 7-18 years. It captures and records continuous raw acceleration data, which will be downloaded in 60-second epochs using ActiLife 6.13.3 software.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Wen Wu, PhD, Principal Investigator — National Taiwan University, College of Medicine
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No